CLINICAL TRIAL: NCT02576145
Title: Immune Response to Neoantigen and Recall Antigen in Pediatric Renal Transplant Recipients Treated With the IL-2R Alfa Monoclonal Antibody, Daclizumab (Zenapax®)
Brief Title: A Study to Assess Immune Response in Pediatric Kidney Transplant Recipients Treated With Daclizumab (Zenapax)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA16215
Record Dates: First submitted 2015-10-05; First posted 2015-10-15 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (With Daclizumab Therapy) (Experimental): Participants who were receiving a full course of 5 doses of daclizumab (1 milligram per kilogram [mg/kg]) with Day 1 vaccine administered immediately prior to the fifth dose.
  Interventions: Biological: DT; Drug: Daclizumab; Biological: KLH
- Group B (Post Daclizumab Therapy) (Active Comparator): Participants who completed a full course of daclizumab therapy in the previous 4 to 18 months.
  Interventions: Biological: DT; Biological: KLH

INTERVENTIONS:
Biological: DT — Diphtheria and Tetanus Toxoid (DT) will be administered intramuscularly as a 1/3 dilution (0.33 flocculation units). The participants will be rechallenged with DT 6 months after Day 29 if failed to show >=1.5 fold increase in lymphocyte proliferative response but have a humoral response.
Drug: Daclizumab — The fifth dose (1 milligram per kilogram [mg/kg]) of daclizumab will be administered in this study to participants who already received four doses (one dose at 1 mg/kg within 24 hours post-transplant and then every other week for 3 doses).
  Other Names: Zenapax
  Arms: Group A (With Daclizumab Therapy)
Biological: KLH — KLH will be administered intradermally with a dose of 250 mcg for participants aged 2 to less than 12 years, and 500 mcg for participants aged 12 to 19 years. The participants will be rechallenged with KLH 6 months after Day 29 if failed to show specified increase in lymphocyte proliferative response or humoral response.

SUMMARY:
This study will assess whether daclizumab impairs the ability of children receiving a kidney transplant to elicit a primary immune response. The anticipated time on study treatment is 1 day, and the target sample size is 82 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Primary renal transplant recipients between 2 and 19 years of age
* Receiving or have received daclizumab in the previous 4-18 months
* Receiving or have received daclizumab less than (<) 24 hours pretransplant and additional courses every other week
* Single organ recipients (kidney only)
* Previous vaccination with tetanus toxoid (TT) prior to transplant
* Receiving a maintenance immunosuppression regimen of a calcineurin inhibitor, mycophenolate mofetil, and prednisone (or equivalent corticosteroid)

Exclusion Criteria:

* Received intravenous gamma globulin or a TT vaccination since transplant
* Experienced rejection within 3 months of receiving study vaccinations and/or treated with lymphocyte preparation or methylprednisolone to reverse suspected acute rejection within 3 months of receiving study vaccinations
* Received any vaccine within 30 days of receiving study vaccinations
* Received plasmapheresis treatment or growth hormone treatment since transplant

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2003-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Los Angeles, California
  - Indianapolis, Indiana
  - Kansas City, Missouri
  - Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (With Daclizumab Therapy): Participants who had a renal transplant prior to 6 weeks of study vaccine administration and who were receiving daclizumab therapy were included. Participants were initially vaccinated with Diphtheria Tetanus Toxoid (DT) vaccine and Keyhole Limpet Hemocyanin (KLH) vaccine at least 30 minutes prior to fifth-dose of daclizumab infusion (i.e. Day 1). The next vaccination with DT and KLH was done on Day 29.
- Group B (Post Daclizumab Therapy): Participants who had a renal transplant and who were within 4 to 18 months of completing daclizumab therapy were included. Participants were vaccinated with Diphtheria Tetanus Toxoid (DT) vaccine and Keyhole Limpet Hemocyanin (KLH) vaccine on Day 1 and Day 29.
Period: Overall Study
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Started | 6 | 5
Completed | 3 | 4
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Acute rejection | 1 | 0
Not completed — Tetanus Titers Decreased | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (5.78) | 12.6 (4.16) | 12.2 (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed a Positive Antibody Response (IgG) to Keyhole Limpet Hemocyanin (KLH) Immunization
Description: Positive antibody response was defined as at least a 2-fold increase in antibody concentration on either Day 43 or Day 57 compared with baseline where baseline was assigned a value of 1 if it was below the limit of quantification. All humoral responses were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 43 or Day 57
Population: All patient population: All participants who were enrolled in the study and received at least 2 vaccine doses and had Day 43 and 57 assessments were included in this population.
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 5 | 5
participants | 2 | 2

2. Secondary Outcome: Number of Participants Who Developed a Positive Cellular Response to KLH Immunization
Description: Positive cellular response was defined as an increase in the 5-bromo-2-deoxyuridine (BrdU) percent total net of at least 1.5-fold compared with baseline, where baseline was assigned a value of 0.5 if <=0, on at least one time point on Days 22, 29, 43 or 57. All cellular responses were assessed by BrdU proliferation assay.
Time Frame: Baseline, Day 22, Day 29, Day 43, and Day 57
Population: All patient population: All participants who were enrolled in the study and received at least 1 vaccine dose were included in this population.
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 2 | 5
participants | 1 | 4

3. Secondary Outcome: Number of Participants Who Developed Both a Positive Antibody Response and a Positive Cellular Response to KLH Immunization
Description: Positive antibody response was defined as at least a 2-fold increase in antibody concentration on either Day 43 or Day 57 compared with baseline where baseline was assigned a value of 1 if it was below the limit of quantification. Positive cellular response was defined as an increase in the 5-bromo-2-deoxyuridine (BrdU) percent total net of at least 1.5-fold compared with baseline, where baseline was assigned a value of 0.5 if <=0, on at least one time point on Days 22, 29, 43 or 57. All humoral responses were assessed by ELISA and all cellular responses were assessed by BrdU proliferation assay.
Time Frame: Baseline, Day 22, Day 29, Day 43 and Day 57
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 2 | 5
participants | 1 | 1

4. Secondary Outcome: Number of Participants Who Developed a Positive Humoral Response to Tetanus Toxoid (TT)
Description: Humoral response to TT was defined as >=1.5 fold increase in antibody concentration from baseline in participants with protective anti-TT IgG level >=0.1 IU/mL. All humoral responses were assessed by ELISA.
Time Frame: Baseline, Day 22, Day 29, Day 43 and Day 57
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 5 | 4
participants | 3 | 3

5. Secondary Outcome: Number of Participants Who Developed a Positive Cellular Response to Tetanus Toxoid (TT)
Description: Positive cellular response was defined as an increase in the BrdU percent total net of at least 1.5-fold compared with baseline, where baseline was assigned a value of 0.5 if <=0, on at least one time point on days 22, 29, 43 or 57. All cellular responses were assessed by BrdU proliferation assay.
Time Frame: Baseline, Day 22, Day 29, Day 43 and Day 57
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 3 | 4
participants | 2 | 3

6. Secondary Outcome: Number of Participants Who Developed a Positive Antibody Response to KLH and Positive Cellular Responses to Both KLH and TT Immunizations
Description: as for outcome 3
Time Frame: Baseline, Day 22, Day 29, Day 43 and Day 57
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 1 | 2
participants | 0 | 1

7. Secondary Outcome: Number of KLH Cellular Nonresponders Who Were Rechallenged and Mounted a Cellular Response to KLH Immunization
Description: Nonresponders (participants who failed to mount cellular responses to KLH) were rechallenged with KLH 6 months after Day 29 (Day 196). For nonresponders, positive cellular response to KLH was defined as an increase in the 5-bromo-2-deoxyuridine (BrdU) percent total net of at least 1.5-fold compared with baseline, where baseline was assigned a value of 0.5 if <=0, on at least one time point up to Day 252. All cellular responses were assessed by BrdU proliferation assay.
Time Frame: Up to Day 252
Population: All patient population: All participants who were enrolled in the study and received at least 2 vaccine doses were included in this population. Only participants who were KLH cellular nonresponders were evaluated.
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

8. Secondary Outcome: Number of Tetanus Cellular Nonresponders Who Were Rechallenged and Mounted a Cellular Tetanus Response
Description: Nonresponders (participants who mount humoral responses but no cellular responses to tetanus vaccination) were rechallenged with TT 6 months after Day 29 (Day 196). For nonresponders, positive cellular response to TT was defined as an increase in the BrdU percent total net of at least 1.5-fold compared with baseline, where baseline was assigned a value of 0.5 if <=0, at any time point up to Day 252. All cellular responses were assessed by BrdU proliferation assay.
Time Frame: up to Day 252
Population: All patient population: All participants who were enrolled in the study and received at least 2 vaccine doses were included in this population. Only participants who were tetanus cellular nonresponders were evaluated.
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

9. Secondary Outcome: Geometric Mean Antibody Concentrations for KLH (IgM and IgG) and TT (IgG)
Description: Due to the small number of participants enrolled in the study, geometric means at Baseline and on Days 22, 29, 43 and 57 were not reported.
Time Frame: Screening, Day 22, Day 29, Day 43 and Day 57
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Percent Expression of 2A3/CD25+ Antibody
Description: CD25 is an antigen that is present on a subset of peripheral blood lymphocytes. The expression of CD25+ on T cell was investigated using antibody 2A3. Blood samples were drawn for evaluation of CD25+ at screening and on Days 29, 57, and 168.
Time Frame: Screening, Day 29, Day 57 and Day 168
Population: All patient population: All participants who were enrolled in the study and received at least 1 vaccine dose were included in this population. Only participants with data available at a particular time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percent expression
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 6 | 5
Percent expression
  Screening, n=1, 5 | 0.10 (NA) — Dispersion is not available as only 1 participant was analysed | 9.44 (3.023)
  Day 29, n=5, 3 | 0.12 (0.084) | 8.53 (2.003)
  Day 57, n=5, 5 | 0.06 (0.055) | 10.18 (2.479)
  Day 168, n=6, 3 | 8.33 (2.670) | 12.53 (4.888)

11. Secondary Outcome: Mean Percent Expression of CD3, CD4, and CD8
Description: Blood samples were obtained for flow activated cell sorter (FACS) analyses of T cell subsets (CD3, CD4, and CD8) on Days 1, 22, 29, 43, and 57. These cells are present on white blood cells and are used as markers to associate cells with immune functions.
Time Frame: Days 1, 22, 29, 43 and 57
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent expression
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 6 | 5
Percent expression
  CD3+, Day 1, n=6, 2 | 76.97 (4.069) | 79.50 (1.414)
  CD3+, Day 22, n=6, 2 | 78.70 (7.211) | 77.25 (1.202)
  CD3+, Day 29, n=5, 2 | 79.82 (9.116) | 78.80 (1.131)
  CD3+, Day 43, n=5, 2 | 76.74 (10.126) | 78.65 (0.778)
  CD3+, Day 57, n=5, 2 | 77.80 (8.460) | 79.20 (3.960)
  CD4+, Day 1, n=6, 2 | 48.87 (7.153) | 36.90 (7.212)
  CD4+, Day 22, n=6, 2 | 48.98 (7.743) | 34.20 (9.051)
  CD4+, Day 29, n=5, 2 | 51.16 (8.830) | 34.85 (7.566)
  CD4+, Day 43, n=5, 2 | 47.08 (8.685) | 34.75 (6.435)
  CD4+, Day 57, n=5, 2 | 47.58 (8.404) | 36.85 (6.718)
  CD8+, Day 1, n=6, 2 | 24.07 (5.452) | 37.30 (9.758)
  CD8+, Day 22, n=6, 2 | 25.15 (6.806) | 38.25 (11.526)
  CD8+, Day 29, n=5, 2 | 24.06 (7.790) | 38.75 (10.394)
  CD8+, Day 43, n=5, 2 | 24.00 (8.405) | 39.00 (8.768)
  CD8+, Day 57, n=5, 2 | 24.86 (7.110) | 38.55 (11.243)

12. Secondary Outcome: Mean Percent Expression of HLA-DR+, CD45RO+ and CD45RA+
Description: Blood samples were obtained for flow activated cell sorter (FACS) analyses of HLA-DR+, CD45RO+ and CD45RA+ on Days 1, 29, and 57. These cells are present on white blood cells and are used as markers to associate cells with immune functions.
Time Frame: Days 1, 29 and 57
Population: All patient population: All participants who were enrolled in the study and received at least 1 vaccine dose were included in this population.Only participants with data available at a particular time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percent expression
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 6 | 5
Percent expression
  HLADR+, Day 1, n=6, 2 | 2.58 (1.098) | 5.80 (3.394)
  HLADR +, Day 29, n=5, 2 | 5.04 (7.720) | 5.10 (4.101)
  HLADR +, Day 57, n=5, 2 | 4.16 (5.126) | 4.55 (3.182)
  CD45RO +, Day 1, n=6, 2 | 22.85 (3.690) | 39.45 (3.889)
  CD45RO +, Day 29, n=5, 2 | 27.04 (4.779) | 39.45 (8.556)
  CD45RO +, Day 57, n=5, 2 | 26.90 (7.027) | 34.45 (3.323)
  CD45RA +, Day 1, n=6, 2 | 69.85 (4.359) | 50.50 (4.384)
  CD45RA +, Day 29, n=5, 2 | 66.86 (5.663) | 52.70 (10.041)
  CD45RA +, Day 57, n=5, 2 | 62.84 (5.999) | 56.15 (5.869)

13. Secondary Outcome: Percentage of Participants With Positive Antibody Response to KLH Immunization at Month 6
Description: Positive antibody response was defined as at least a 2-fold increase in antibody concentration on Month 6 compared with baseline where baseline was assigned a value of 1 if it was below the limit of quantification. All humoral responses were assessed by enzyme-linked immunosorbent assay (ELISA). Due to the small number of participants enrolled in the study, percentage of participants with positive antibody response to KLH immunization at Month 6 was not reported.
Time Frame: Month 6
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of KLH Antibody Nonresponders Who Underwent Rechallenge and Mounted a KLH Antibody Response
Description: Nonresponders (participants who failed to mount antibody responses to KLH) were rechallenged with KLH 6 months after Day 29 (Day 196). For nonresponders, positive antibody response to KLH was defined as at least a 2-fold increase in antibody concentration at any time point up to Day 252 compared with baseline where baseline was assigned a value of 1 if it was below the limit of quantification. All humoral responses were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Up to Day 252
Population: All patient population: All participants who were enrolled in the study and received at least 2 vaccine doses were included in this population. Only participants who were KLH Antibody nonresponders were evaluated.
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 2 | 1
participants | 1 | 1

15. Secondary Outcome: Number of Participants With a Positive Delayed Type Hypersensitivity (DTH) Response After KLH Immunization
Description: DTH skin reactions were assessed 48 hours after each KLH immunization given on Day 1 and on Day 29. A positive response was defined as an induration >=5 mm.
Time Frame: Day 1 and Day 29
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 6 | 5
participants | 0 | 1

16. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes
Time Frame: Up to Month 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Number analyzed (Participants) | 6 | 5
participants
  Any AE | 6 | 4
  Any SAE | 3 | 2

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: SAEs and AEs were collected in members of All Patient Population, comprised of all participants who were enrolled in the study and received at least 1 vaccine dose.
Arm/Group | Group A (With Daclizumab Therapy) | Group B (Post Daclizumab Therapy)
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (With Daclizumab Therapy) (N=6) | Group B (Post Daclizumab Therapy) (N=5)
BK virus infection (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (With Daclizumab Therapy) (N=6) | Group B (Post Daclizumab Therapy) (N=5)
Hordeolum (Infections and infestations) | 1 | 0
Upper respiratory tract Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Urinary sediment present (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Injection site induration (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.